CLINICAL TRIAL: NCT05619627
Title: Utility of Oral Dexmedetomidine as the Sole Sedative Agent in Pediatric Population Undergoing MRI
Brief Title: Oral Dexmedetomidine in Pediatric MRI
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Soroush Merchant (Other)
Responsible Party: Sponsor-Investigator, Soroush Merchant, Director of Medical Pain Service, Principal Investigator, Assistant Professor of Anesthesiology, MD, MS, Children's Mercy Hospital Kansas City
Organization: Children's Mercy Hospital Kansas City (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00002526
Record Dates: First submitted 2022-10-05; First posted 2022-11-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Anesthesia
Keywords: Oral dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Anesthesia, General; Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective Pilot Study, Single-site, open-label, phase I dose escalation trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Dexmedetomidine 4 mcg/kg (Experimental): Group One: Subjects will receive oral dexmedetomidine 4 mcg/kg 2 hours prior to MRI
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 6 mcg/kg (Experimental): Group Two: Subjects will receive oral dexmedetomidine 6 mcg/kg 2 hours prior to MRI
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 8 mcg/kg (Experimental): Group Three: Subjects will receive oral dexmedetomidine 8 mcg/kg 2 hours prior to MRI
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 10 mcg/kg (Experimental): Group Four: Subjects will receive oral dexmedetomidine 10 mcg/kg 2 hours prior to MRI
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 12 mcg/kg (Experimental): Group Five: Subjects will receive oral dexmedetomidine 12 mcg/kg 2 hours prior to MRI
  Interventions: Drug: Dexmedetomidine
- General anesthesia (Active Comparator): Control group: Subjects will receive general anesthesia for their MRI
  Interventions: Drug: General Anesthesia (control group)

INTERVENTIONS:
Drug: Dexmedetomidine — Participants will receive oral dexmedetomidine as the sole sedative agent for undergoing MRI
  Arms: Dexmedetomidine 10 mcg/kg; Dexmedetomidine 12 mcg/kg; Dexmedetomidine 4 mcg/kg; Dexmedetomidine 6 mcg/kg; Dexmedetomidine 8 mcg/kg
Drug: General Anesthesia (control group) — Participants will receive general anesthesia for their MRI
  Arms: General anesthesia

SUMMARY:
The objective of this preliminary study is to assess the utility of oral dexmedetomidine as the sole sedative agent in pediatric population undergoing MRI.

DETAILED DESCRIPTION:
MRI is an important and robust medical imaging technique that has become the cornerstone for radiologic studies. Superior image quality and resolution especially for soft tissue imaging, without the use of ionizing radiation, has made MRI a dominant imaging modality in pediatrics. Despite its many advantages, MRI is not child friendly. Lengthy scan times, the need for lying motionless in a confined space, excessive noise and vibration during image acquisition, are all factors that have made anesthesia an integral part of pediatric MRI.

General anesthesia is a state of medically induced unconsciousness, analgesia and muscle relaxation which is required for most invasive medical procedures. Despite being painless, MRI scans are highly susceptible to motion artifact and require a state of immobility that may not be obtainable in awake uncooperative children. While very safe, general anesthesia carries potential risk of serious morbidity and mortality secondary to aspiration during instrumentation of the airway, hypoxia and hypoventilation secondary to laryngospasm/bronchospasm and hemodynamic instability. Therefore, sedation may be an appropriate technique to offer anxiolysis, amnesia and immobility while maintaining airway reflexes with limited impact on ventilation and hemodynamics for non-stimulating procedures such as imaging. Aside from having a more favorable risk/benefit profile as compared to general anesthesia when it comes to radiologic studies, sedation is also less costly and burdensome on anesthesia departments and could provide immense cost-saving measures for healthcare institutions at large.

While there are many intravenous (IV) sedatives, establishing IV access while awake could be very traumatizing, leaving a lasting negative impression of the healthcare environment in a child's mind. Hence, enteral medications may be more acceptable and child friendly. This is especially valuable in patients who require repeated surveillance imaging and who demonstrate heightened level of anxiety and fear with each visit. Among sedative agents that could be administered enterally, dexmedetomidine may be superior due to minimal respiratory depression while providing anxiolysis and analgesia. Of note, dexmedetomidine is a highly selective alpha2-adrenoreceptor agonist that exerts its hypnotic action through activation of central pre- and postsynaptic alpha2-receptors in the locus coeruleus, mimicking natural sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Participants 3-6 years old, male and female, all races and ethnicities
2. Requiring a clinically indicated MRI with general anesthesia

Exclusion Criteria:

1. Refusal to take oral dexmedetomidine
2. Known allergy to dexmedetomidine
3. Inability to take dexmedetomidine at least 90 minutes prior to start of the MRI
4. Medical contraindications to administration of dexmedetomidine including:

   1. Unstable cardiac status including life threatening arrhythmias, abnormal cardiac anatomy, significant cardiac dysfunction
   2. Current use of digoxin
   3. Moya Moya disease
   4. New onset stroke
5. American Society of Anesthesiologists (ASA) physical status classification > II
6. Contraindications to administering sedation including:

   1. Active and uncontrolled gastroesophageal reflux
   2. Active and uncontrolled vomiting
   3. Current or recent history of apnea
   4. Active respiratory disease including pneumonia, bronchitis, respiratory syncytial virus infection, asthma exacerbation
   5. Craniofacial anomalies
7. Inability to have MRI scans
8. Non-English speaking volunteers

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Oral dexmedetomidine dose with adverse event below moderate risk, as designated by SIVA, to obtain adequate MRI study | From date of the first enrollment until the end of assessment of data collected from the last participant, up to 70 weeks
  The primary outcome is determining a dose of oral dexmedetomidine that will safely (adverse event (AE) below moderate risk, as designated by the World Society of Intravenous Anesthesia (SIVA) adverse sedation event reporting tool) provide adequate sedation to successfully complete an MRI. Images should have adequate quality and resolution to be interpretated and will be graded by an attending radiologist. Each MRI sequence will be graded 1-3. 1: no-mild motion artifact; 2: moderate motion artifact; 3: severe motion artifact (non-diagnostic).

CONTACTS AND LOCATIONS:
Overall Officials: Soroush Merchant, MD, MS, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication

REFERENCES:
- [Background] Mason KP, Roback MG, Chrisp D, Sturzenbaum N, Freeman L, Gozal D, Vellani F, Cavanaugh D, Green SM. Results from the Adverse Event Sedation Reporting Tool: A Global Anthology of 7952 Records Derived from >160,000 Procedural Sedation Encounters. J Clin Med. 2019 Dec 1;8(12):2087. doi: 10.3390/jcm8122087. PMID 31805686
- [Background] Mason KP, Green SM, Piacevoli Q; International Sedation Task Force. Adverse event reporting tool to standardize the reporting and tracking of adverse events during procedural sedation: a consensus document from the World SIVA International Sedation Task Force. Br J Anaesth. 2012 Jan;108(1):13-20. doi: 10.1093/bja/aer407. PMID 22157446
- [Background] Sajid B, Mohamed T, Jumaila M. A comparison of oral dexmedetomidine and oral midazolam as premedicants in children. J Anaesthesiol Clin Pharmacol. 2019 Jan-Mar;35(1):36-40. doi: 10.4103/joacp.JOACP_20_18. PMID 31057237
- [Background] Weerink MAS, Struys MMRF, Hannivoort LN, Barends CRM, Absalom AR, Colin P. Clinical Pharmacokinetics and Pharmacodynamics of Dexmedetomidine. Clin Pharmacokinet. 2017 Aug;56(8):893-913. doi: 10.1007/s40262-017-0507-7. PMID 28105598
- [Background] Anttila M, Penttila J, Helminen A, Vuorilehto L, Scheinin H. Bioavailability of dexmedetomidine after extravascular doses in healthy subjects. Br J Clin Pharmacol. 2003 Dec;56(6):691-3. doi: 10.1046/j.1365-2125.2003.01944.x. PMID 14616431
- [Background] Mason KP, Zurakowski D, Zgleszewski SE, Robson CD, Carrier M, Hickey PR, Dinardo JA. High dose dexmedetomidine as the sole sedative for pediatric MRI. Paediatr Anaesth. 2008 May;18(5):403-11. doi: 10.1111/j.1460-9592.2008.02468.x. Epub 2008 Mar 18. PMID 18363626
- [Background] Lin L, Guo X, Zhang MZ, Qu CJ, Sun Y, Bai J. Pharmacokinetics of dexmedetomidine in Chinese post-surgical intensive care unit patients. Acta Anaesthesiol Scand. 2011 Mar;55(3):359-67. doi: 10.1111/j.1399-6576.2010.02392.x. PMID 21288220
- [Background] Iirola T, Ihmsen H, Laitio R, Kentala E, Aantaa R, Kurvinen JP, Scheinin M, Schwilden H, Schuttler J, Olkkola KT. Population pharmacokinetics of dexmedetomidine during long-term sedation in intensive care patients. Br J Anaesth. 2012 Mar;108(3):460-8. doi: 10.1093/bja/aer441. Epub 2012 Jan 25. PMID 22277665
- [Background] Lee S, Kim BH, Lim K, Stalker D, Wisemandle W, Shin SG, Jang IJ, Yu KS. Pharmacokinetics and pharmacodynamics of intravenous dexmedetomidine in healthy Korean subjects. J Clin Pharm Ther. 2012 Dec;37(6):698-703. doi: 10.1111/j.1365-2710.2012.01357.x. Epub 2012 May 31. PMID 22650799
- [Background] Hannivoort LN, Eleveld DJ, Proost JH, Reyntjens KM, Absalom AR, Vereecke HE, Struys MM. Development of an Optimized Pharmacokinetic Model of Dexmedetomidine Using Target-controlled Infusion in Healthy Volunteers. Anesthesiology. 2015 Aug;123(2):357-67. doi: 10.1097/ALN.0000000000000740. PMID 26068206
- [Background] Potts AL, Anderson BJ, Warman GR, Lerman J, Diaz SM, Vilo S. Dexmedetomidine pharmacokinetics in pediatric intensive care--a pooled analysis. Paediatr Anaesth. 2009 Nov;19(11):1119-29. doi: 10.1111/j.1460-9592.2009.03133.x. Epub 2009 Aug 25. PMID 19708909
- [Background] Chamadia S, Pedemonte JC, Hobbs LE, Deng H, Nguyen S, Cortinez LI, Akeju O. A Pharmacokinetic and Pharmacodynamic Study of Oral Dexmedetomidine. Anesthesiology. 2020 Dec 1;133(6):1223-1233. doi: 10.1097/ALN.0000000000003568. PMID 32986820
- [Background] Dashiff CJ, Weaver M. Development and testing of a scale to measure separation anxiety of parents of adolescents. J Nurs Meas. 2008;16(1):61-80. doi: 10.1891/1061-3749.16.1.61. PMID 18578110
- [Background] Keles S, Kocaturk O. Comparison of oral dexmedetomidine and midazolam for premedication and emergence delirium in children after dental procedures under general anesthesia: a retrospective study. Drug Des Devel Ther. 2018 Mar 28;12:647-653. doi: 10.2147/DDDT.S163828. eCollection 2018. PMID 29636599
- [Background] Weldon BC, Watcha MF, White PF. Oral midazolam in children: effect of time and adjunctive therapy. Anesth Analg. 1992 Jul;75(1):51-5. doi: 10.1213/00000539-199207000-00010. PMID 1616162
- [Background] Shukry M, Clyde MC, Kalarickal PL, Ramadhyani U. Does dexmedetomidine prevent emergence delirium in children after sevoflurane-based general anesthesia? Paediatr Anaesth. 2005 Dec;15(12):1098-104. doi: 10.1111/j.1460-9592.2005.01660.x. PMID 16324031